CLINICAL TRIAL: NCT06654804
Title: Contrast-Enhanced Ultrasound Biomarker for Prognostication and Guidance of Surgical Treatment in Acute Traumatic Spinal Cord Injury
Brief Title: Contrast-enhanced Ultrasound in the Treatment of Acute Spinal Cord Injury
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Christoph Hofstetter, Associate Professor: Neurological Surgery, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00017544
Record Dates: First submitted 2024-05-26; First posted 2024-10-23 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Acute Spinal Cord Injury
MeSH Terms: interventions — perflutren

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Contrast-enhanced ultrasound in traumatic spinal cord injury (Experimental): A bolus IV injection of Perflutren lipid contrast agent will be given. Continuous imaging will be obtained.
  Interventions: Drug: Perflutren lipid

INTERVENTIONS:
Drug: Perflutren lipid — Bolus injection of contrast during spinal decompression surgery for the treatment of traumatic spinal cord injury. Ultrasound imaging will then be used to collect images of the spinal cord injury to record perfusion, inflow and washout.
  Other Names: Definity

SUMMARY:
Patients with traumatic spinal cord injury (tSCI) often suffer from spinal cord swelling inside the thecal sac, which contains the spinal cord and surrounding fluid, leading to increased pressure on the spinal cord tissue and decreased spinal cord blood flow at the site of injury. The combination of increased pressure and decreased blood flow causes vascular hypoperfusion of the spinal cord and exacerbates the severity of injury. This is also referred to as secondary injury. Thus, knowledge of spinal cord hypoperfusion would allow the treating physician to optimize the hemodynamic condition of the patient with acute spinal cord injury and potentially improve functional outcomes.

DETAILED DESCRIPTION:
The investigators plan to use contrast-enhanced ultrasound (CEUS) to determine a decrease in the blood flow in the spinal cord at the site of injury, during the routine surgery that these patients require to decompress and stabilize their injured spine. This may help the investigators to determine the efficacy of certain treatments in improving blood flow and patients suffering from traumatic spinal cord injury.

Patients presenting to Harborview Medical Center with a diagnosis of traumatic spinal cord injury will be screened for participation. Many of these patients require emergent or urgent surgery for decompression of the spinal cord and stabilization of the spine.

The patient will be taken to the operating room as per routine. After completion of the key elements of surgery, namely posterior decompression, and stabilization of the cervical or thoracic spinal cord, CEUS will be performed. Importantly, the proposed trial does not prolong the time before surgical decompression and stabilization are accomplished. Moreover, it does not increase the invasiveness of the procedure as it is collected at the final stage of the routine procedure. A hand-held intraoperative ultrasound probe will be used to collect sagittal images of the spinal cord centered above the spinal cord injury. A bolus IV injection of the contrast agent will be given. Continuous imaging will be obtained to record contrast inflow and washout.

Post-operatively, the participant will receive routine MRI imaging within one week (health status permitting) and one year.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age minimum
* Acute spinal cord injury fpr less than 24 hours
* Injury ranging from mild spinal cord injury where motor function is preserved (AIS A) to complete injury where there is no motor or sensory function below the leel of the injury (AIS D)
* Medically stable to undergo routine dorsal decompression, spinal realignment
* and stabilizing with segmental instrumentation

Exclusion Criteria:

* Younger than 18 years old
* Neurological lower extremity exam missing or intact
* Traumatic head injury with a Glasgow score of 11 or lower
* Cord injury level caudal to T10 (thoracic spine level 10)
* A known sensitivity to lipid microsphere or its components, such as polyethylene glycol (PEG)
* A history of anaphylactoid reactions from ultrasound enhancing agents
* A known history of cardiopulmonary conditions
* Cardiac shunt

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-09-28 (Actual); Primary Completion 2027-09-15 (Estimated); Study Completion 2027-09-15 (Estimated)

PRIMARY OUTCOMES:
Outcomes of all subjects who received contrast enhanced ultrasound imaging, to check perfusion during the surgical repair of an acute spinal cord injury. | Two years
  Knowledge of spinal cord hypoperfusion will allow the physician to optimize the hemodynamic condition of acute spinal cord injury and potentially improve outcomes. The investigators plan to use contrast-enhanced ultrasound to determine decreased blood flow in the spinal cord at the site of injury, during the routine surgery that these patients require to decompress and stabilize their injured spine.

SECONDARY OUTCOMES:
Determine the prognostic capacity of CEUS biomarker for acute tSCI and surgical outcomes/recovery in spine injury/surgery. | Two years
  Measure the outcomes of spinal cord decompression surgery in patient population.
  The protocol is designed to develop a standardized operating procedure for prognostic intraoperative biomarker acquisition and readout. Inter- and intra-rater reliability will be scored, and the CEUS markers will be validated with tSCI severity reference standards such as MRI biomarkers and AIS score. Aim 2 of the study will also focus on determining the prognostic capacity for chronic neurological outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Hofstetter, MD, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington Harborview Medical Center, Seattle, Washington, United States